CLINICAL TRIAL: NCT02204813
Title: To Define the Role of GLP-1 for Improving Glucose Homeostasis in Humans Following Gastric Bypass Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 08-0861F; R01DK088126 (NIH)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Bypass, Gastric; Roux-en-Y Gastric Bypass; Vertical Sleeve Gastrectomy; Gastric Banding; Bariatric Surgery
Keywords: Gastric Bypass; RYGB; GLP-1; Xenin; Insulin Secretion; Glucose Homeostasis; Vertical Sleeve; Lap Band
MeSH Terms: interventions — Albumins

STUDY DESIGN:
Intervention Model Description: Patients with prior RYGB surgery receive all interventions, each on a separate day.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Post RYGB Surgery (Experimental): Healthy, weight stable individuals, with previous Roux-en-Y gastric bypass surgery. No clinical evidence of type 2 diabetes before and after surgery. Each participant will receive placebo or the indicated doses of xenin-25.
  Interventions: Drug: Placebo; Drug: Lo-Xenin; Drug: Hi-Xenin; Drug: Extra Hi-Xenin

INTERVENTIONS:
Drug: Placebo — A liquid mixed meal containing 1.5 grams of acetaminophen will be ingested in 7 equal portions from 0-30 minutes.
  Starting at minus 15 minutes, an intravenous infusion of albumin alone (placebo) will be administered for 5.25 hours.
  Other Names: Control; Albumin Alone
Drug: Lo-Xenin — A liquid mixed meal containing 1.5 grams of acetaminophen will be ingested in 7 equal portions from 0-30 minutes.
  Starting at minus 15 minutes, an intravenous infusion of xenin-25 at a dose of 4 pmoles/kg/min will be administered for 5.25 hours.
  Other Names: Lo-Xen
Drug: Hi-Xenin — A liquid mixed meal containing 1.5 grams of acetaminophen will be ingested in 7 equal portions from 0-30 minutes.
  Starting at minus 15 minutes, an intravenous infusion of xenin-25 at a dose of 12 pmoles/kg/min will be administered for 5.25 hours.
  Other Names: Hi-Xen
Drug: Extra Hi-Xenin — A liquid mixed meal containing 1.5 grams of acetaminophen will be ingested in 7 equal portions from 0-30 minutes.
  Starting at minus 15 minutes, an intravenous infusion of xenin-25 at a dose of 24 pmoles/kg/min will be administered for 5.25 hours.
  Other Names: XHi-Xen

SUMMARY:
There is a marked and long-lasting improvement in glucose homeostasis that follows Roux-en-y gastric bypass surgery (RYGB) in humans. This improvement has been attributed in large part to an intestinal hormone, called GLP-1, that is released into the circulation immediately after eating. The purpose of this study is to determine if GLP-1 mediates the beneficial effects of RYGB surgery on glucose homeostasis in humans.

DETAILED DESCRIPTION:
To conduct this study, we will enroll humans who previously underwent Roux-en-Y gastric bypass surgery, who are medically and weight stable and with no signs of type 2 diabetes either before or after surgery. Potential subjects will first be screened for eligibility and also to verify that they can safely participate in the study. Each study subject will be administered a meal tolerance test (MTT) on 3 separate occasions. For the MTT, a liquid meal (Boost Plus) will be ingested following an overnight fast. A primed-continuous infusion of vehicle alone (human albumin) or xenin-25 alone (at a dose of 4 or 12 pmoles x kg-1 x min-1) will be initiated 15 minutes before the meal is ingested. Blood samples will be collected before and during the MTT for the measurement of glucose and insulin levels, as well as a host of other hormones. A comparison of the results will tell us if the effects of xenin-25 on insulin release are mediated by GLP-1 in humans.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be able to consent for their own participation (no mental impairment affecting cognition or willingness to follow study instructions).
* Healthy, weight stable, with previous Roux-en-Y gastric bypass surgery and no clinical evidence of type 2 diabetes either before and after Roux-en-Y gastric bypass surgery.
* Women of childbearing potential must be currently taking/using a method of birth control that is acceptable to the investigators. A pregnancy test will be done at the beginning of each visit. Any woman with a positive pregnancy test will be removed from the study.
* Willingness to return have 8-10ml of blood drawn 25-30 days after the last Xenin infusion; to check for Xenin peptide antibodies that MAY develop. (All efforts will be made to complete this visit during study participation.)

Exclusion Criteria:

* Lacks cognitive ability to sign the consent &/or follow the study directions for themselves.
* Women unwilling to comply with using an acceptable method of contraception during the course of the study, or who are currently breast-feeding.
* Volunteers with a history of Acute Pancreatitis.
* Volunteers with a history of cancer (except for skin cancer).
* Volunteer with a history of Chronic Pancreatitis and/or risk factors for chronic pancreatitis including hypertriglyceridemia (triglycerides >400mg/ml) hypercalcemia (blood calcium level >11.md/dl) and/or the presence of gallstones.
* Subjects taking medications known to affect glucose tolerance.
* Hematocrit from the lab is below 33% (or if the finger stick hemoglobin measured with the HemoCue 201+ is <11.2 g/dl).
* Any major medical conditions, or conditions that in the opinion of the PI make the subject unsuitable for the study.
* Subjects with abnormal kidney function as measured by the Creatinine concentration will be excluded.
* Subjects with a history of active liver disease or AST/ALT levels >2X upper limit of normal will also be excluded.
* Total Bilirubin levels should be <2.
* Subjects unwilling to allow the use of their own blood or albumin in the preparation of the peptides. (The blood will prevent sticking of the peptide to the tubing; an alternative method has been sought but not found.)
* Unwillingness to return have 8-10ml of blood drawn 25-30 days after the last Xenin infusion; to check for Xenin peptide antibodies that MAY develop. (All efforts will be made to complete this visit during study participation.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2015-11-17 (Actual)

PRIMARY OUTCOMES:
Insulin secretion rates (ISRs) during each treatment | 5.5 hours
  ISRs will be measured at various times before and after ingestion of a liquid mixed meal.

SECONDARY OUTCOMES:
Plasma glucose levels during each treatment. | 5.5 hours
  Plasma glucose levels will be measured at various times before and after ingestion of a liquid mixed meal.
Plasma glucagon levels during each treatment. | 5.5 hours
  Plasma glucagon levels will be measured at various times before and after ingestion of a liquid mixed meal.
Plasma GLP-1 during each treatment. | 5.5 hours
  Plasma GLP-1 levels will be measured at various times before and after ingestion of a liquid mixed meal.
Plasma C-peptide levels during each treatment. | 5.5 hours
  Plasma C-peptide levels will be measured at various times before and after ingestion of a liquid mixed meal.
The rate of gastric emptying during each treatment. | 5.5 hours
  The rate of gastric emptying will be estimated after ingestion of a liquid mixed meal.

CONTACTS AND LOCATIONS:
Overall Officials: Burton M Wice, PhD, Principal Investigator — Washington University School of Medicine; Dominic Reeds, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sterl K, Wang S, Oestricker L, Wallendorf MJ, Patterson BW, Reeds DN, Wice BM. Metabolic responses to xenin-25 are altered in humans with Roux-en-Y gastric bypass surgery. Peptides. 2016 Aug;82:76-84. doi: 10.1016/j.peptides.2016.06.001. Epub 2016 Jun 7. PMID 27288245